CLINICAL TRIAL: NCT06374745
Title: An Integrated Algorithm for Surgical Intervention in Chronic Lymphedema After Breast Cancer Treatment: The Basel Lymphedema Protocol
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Sana Kliniken Düsseldorf GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-01307; mu24Kappos
Record Dates: First submitted 2024-04-10; First posted 2024-04-19 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Lymphedema; Breast Cancer
Keywords: Post-surgical Treatment; Chronic Lymphedema Treatment
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the investigators is to develop an integrated algorithm for surgical treatment of chronic lymphedema after breast cancer surgery. This will be achieved by retrospectively analysing a subgroup of patients who had breast cancer-related surgery prior to lymphedema.

DETAILED DESCRIPTION:
Evidence-based surgical treatment recommendations for lymphedema post breast cancer surgery are practically non-existent. In fact, the meager literature on this matter takes into account only quality of life or patient reported outcome - if at all. In light of the heavy burden imposed upon a large portion of breast cancer survivors by chronic lymphedema, the investigators' study aims to create an evidence-based treatment protocol - "The Basel Lymphedema Protocol" - to guide surgeons in taking the best course of action when advising patients, engaging in shared-decision and performing surgery to reduce lymphedema post breast cancer treatment. Accordingly, one of the investigators' driving goals is to allow surgeons to one day be able consistently rely on hard data.

This study is ultimately based on the investigators' intent to further patient welfare. To this effect, creating an integrated algorithm based on concrete, tangible data will not only aid patients by leading to improved treatment of their chronic lymphedema and enabling higher quality of life, but it will also bolster access to adequate coverage. For at present, surgical treatment of lymphedema requires submitting a request for a commitment to cover costs to health insurance providers. This is a protracted, tedious and - unfortunately - an oftentimes fruitless endeavour. However, by having a strong factual basis - more scientific data and peer-reviewed studies - such requests gain a much greater chance of success. To this end, the current study certainly has the capacity to pave the way and set evidence-based standards. And lastly, the creation and implementation of "The Basel Lymphedema Protocol" would strongly reflect the tenets and purpose of personalized/precision medicine - treatment tailored to the unique patient - and by so doing, refine resource allocation and cost-effectiveness of the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* status post breast cancer or status post another type of cancer or status post no cancer
* chronic lymphedema - lymphedema lasting over three months - present prior to surgical treatment
* one type of surgical procedure for treatment of chronic lymphedema or a combination of surgical procedures for treatment of chronic lymphedema was performed
* one or any combination of the following surgical procedures was used in each individual patient: Lymph Node-Vein Anastomosis (LNVA) , Lymphaticovenous Anastomosis (LVA), Tumescent Liposuction (TL), Vascularized Lymph Node Transfer (VLNT) and/or Water-Assisted Liposuction (WAL)

Exclusion Criteria:

* inclusion criteria not met
* loss to follow-up (data not successfully collected)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with lymphedema surgery performed at the University Hospital Basel between 2015 and 2023.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-01-02 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
To design an integrated algorithm for surgical treatment of chronic lymphedema after breast cancer surgery. | baseline to follow up (no later than December 2024)
  To design an integrated algorithm for surgical treatment of chronic cancer-associated lymphedema using the following variables captured in Primary Outcomes 2 to 21.
Date of follow-up procedure | baseline to follow up (no later than December 2024)
  Date of follow-up procedure.
Follow-up and type of lymphedema surgery | baseline to follow up (no later than December 2024)
  If applicable, follow-up and type of lymphedema surgery
Circumferences of the affected and unaffected side | baseline to follow up (no later than December 2024)
  Circumferences of the affected and unaffected side preoperatively and at postoperative time points.
Postoperative complications | baseline to follow up (no later than December 2024)
  Postoperative complications
Surgery duration. | baseline to follow up (no later than December 2024)
  Surgery duration in minutes.
Type of lymphedema surgery | baseline to follow up (no later than December 2024)
  Type of lymphedema surgery including number of anastomoses, localization, long-term patency.
Date of lymphedema surgery | baseline to follow up (no later than December 2024)
  Date of lymphedema surgery.
Use of compression stockings | baseline to follow up (no later than December 2024)
  Use of compression stockings
Number of lymphedema drainages per week | baseline to follow up (no later than December 2024)
  Number of lymphedema drainages per week.
Stage of lymphedema | baseline to follow up (no later than December 2024)
  Stage of lymphedema (stage I, II or III)
Duration of lymphedema | baseline to follow up (no later than December 2024)
  Duration of lymphedema.
Location of lymphedema | baseline to follow up (no later than December 2024)
  Location of lymphedema.
Subsequent cancer treatment | baseline to follow up (no later than December 2024)
  Subsequent cancer treatment (Chemotherapy, Radiotherapy)
Date of cancer related surgery | baseline to follow up (no later than December 2024)
  Date of cancer related surgery
Tumor staging | baseline to follow up (no later than December 2024)
  Tumor staging, considering the following parameters: tumor node metastasis (TNM), resection status of the cancerous growth (R), lymphatic vessel invasion by cancerous cells (L), venous invasion by cancerous cells (V) and grade of cancer cells (G).
Tumor location | baseline to follow up (no later than December 2024)
  Tumor location (right, left, both sides).
BMI | baseline to follow up (no later than December 2024)
  Patient's BMI in kg/m2.
Comorbidities | baseline to follow up (no later than December 2024)
  Existence of comorbidities.
Age | baseline to follow up (no later than December 2024)
  Patient's age in years.
Gender | baseline to follow up (no later than December 2024)
  Patient's gender, given the possibilities male or female.

SECONDARY OUTCOMES:
Analysis of cohort subgroups: all patients who had surgery related to any kind of cancer prior to their lymphedema | baseline to follow up (no later than December 2024)
  Analysis of cohort subgroups: all patients who had surgery related to any kind of cancer prior to their lymphedema
Analysis of cohort subgroups: all patients who had surgery related to a specific kind of cancer prior to their lymphedema, e.g. vulvar, cervical or uterine cancer | baseline to follow up (no later than December 2024)
  Analysis of cohort subgroups: all patients who had surgery related to a specific kind of cancer prior to their lymphedema, e.g. vulvar, cervical or uterine cancer
Analysis of cohort subgroups: all patients who had no history of cancer and thus no cancer-related surgery in their medical history | baseline to follow up (no later than December 2024)
  Analysis of cohort subgroups: all patients who had no history of cancer and thus no cancer-related surgery in their medical history
Analysis of cohort subgroups: all patients with chronic lymphedema regardless of whether or not they have an oncological history | baseline to follow up (no later than December 2024)
  Analysis of cohort subgroups: all patients with chronic lymphedema regardless of whether or not they have an oncological history
Analysis of cohort subgroups: all patients who underwent DIEP flap or TRAM flap or LDM flap or implant based breast reconstruction or BCS | baseline to follow up (no later than December 2024)
  Analysis of cohort subgroups: all patients who underwent Deep Inferior Epigastric Perforator (DIEP) flap or Transverse Rectus Abdominis Myocutaneous (TRAM) flap or Latissimus Dorsi Myocutaneous (LDM) flap or implant based breast reconstruction or Breast Conserving Surgery (BCS)
Analysis of cohort subgroups: exploratory | baseline to follow up (no later than December 2024)
  Analysis of cohort subgroups: exploratory

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth A Kappos, PD Dr. med, Principal Investigator — USB
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided